CLINICAL TRIAL: NCT01973816
Title: Randomized Trial Comparing Functional Digestive Outcomes Related to Two Types of Management of Rectal Endometriosis: Continuous Hormonal Treatment and Curative Surgery
Brief Title: MEdical Versus SUrgical Treatments of Rectal Endometriosis
Acronym: MESURE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 2013/001/HP
Record Dates: First submitted 2013-10-25; First posted 2013-11-01 (Estimated); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Endometriosis
Keywords: deep endometriosis;; rectal endometriosis;; rectal shaving;; colorectal resection;; bowel endometriosis
MeSH Terms: conditions — Endometriosis | interventions — Estradiol; Administration, Cutaneous; Cyproterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Medical treatment (Experimental): The patients received triptoreline and add back therapy by estradiol during 6 months, followed by daily intake of cyproterone acetate and add back therapy during 18 months.
  Interventions: Drug: Triptoreline 11.25 i.v.; Estradiol 0.5% percutaneous gel;; Drug: Cyproterone acetate 50 mg; estradiol 0.5% percutaneous
- Surgical (Active Comparator): The patients are managed by rectal surgery (depending on the surgeon choice: rectal shaving, rectal disc excision or colorectal resection) followed by the prevention of recurrences by daily intake of cyproterone acetate and add back therapy during 18 months.
  Interventions: Procedure: rectal shaving; rectal disc excision; colorectal resection; Drug: Estradiol 0.5% percutaneous gel; Cyproterone acetate 50 mg oral

INTERVENTIONS:
Drug: Triptoreline 11.25 i.v.; Estradiol 0.5% percutaneous gel; — Triptoreline 11.25 administered for 3 months, two consecutive cures Estradiol administered daily for 6 months
  Arms: Medical treatment
Procedure: rectal shaving; rectal disc excision; colorectal resection
  Arms: Surgical
Drug: Cyproterone acetate 50 mg; estradiol 0.5% percutaneous — Daily intake for 18 months
  Arms: Medical treatment
Drug: Estradiol 0.5% percutaneous gel; Cyproterone acetate 50 mg oral — Daily intake during 24 months
  Arms: Surgical

SUMMARY:
The purpose of this study is to determine whether, in women with deep endometriosis involving the rectum and not intending to get pregnant, continuous hormonal treatment would be followed by better digestive functional outcomes than curative rectal surgery. Are included women from 35 to 50 years presenting with deep endometriosis infiltrating at least the muscular layer of the rectum and not having pregnancy intention.

The main outcome concerns the quality of digestive function 24 after the onset of the treatment, assessed using a composite variable: patient considering that digestive function is normal AND the Knowles-Eccersley-Scott-Symptom Questionnaire (KESS score) <7 AND the Gastrointestinal Quality of Life Index (GIQLI) score >100.

Secondary outcomes are: presence of severe constipation, increased frequency of daily bowel movements, anal incontinence, postoperative dysuria, Biberoglou & Behrman score, quality of life SF36 score, KESS score, GIQLI, Wexner score of anal continence, Bristol stools score, the rate of postoperative complications, medical treatment adverse outcomes, the rate of additional endoscopic and surgical procedures.

The randomization is central, once the physician asses the diagnosis, explain the study's principle and rece In the arm A, the patients received triptoreline and add back therapy by estradiol during 6 months, followed by daily intake of cyproterone acetate and add back therapy during 18 months.

In the arm B, patients are managed by rectal surgery (depending on the surgeon choice: rectal shaving, rectal disc excision or colorectal resection) followed by the prevention of recurrences by daily intake of cyproterone acetate and add back therapy during 18 months.

The number of subjects required is 78 (39 on each arm). Inclusions period is estimated at 24 months. The length of the follow up is 24 months. The patients have 8 visits in the arm A, and 7 visits in the arm B.

Eleven French tertiary referral centres will enrol patients in the trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 35-50
* No menopause
* Digestive complaints: defecation pain, dyskesia, diarrhea, constipation, rectorrhage
* Imaging assessment revealing deep endometriosis involving at least the muscular rectal layer
* No intention to get pregnant during the following 24 months
* Negative urinary pregnancy test
* Affiliated to the French Social Security System

Exclusion Criteria:

* Pregnant women or during the breastfeeding
* Pregnancy intention or lack of efficient contraception
* Unexpected rectal endometriosis intraoperatively revealed
* Refus of one of treatments planned in the two arms
* Severe disease requiring surgical treatment in emergency (bowel occlusion, ureteral stenosis or hydronephrosis), severe dyspareunia
* Contraindications to hormonal treatment or surgery
* Major thromboembolic factors
* Antecedents of inflammatory bowel diseases, cancer or colorectal resection
* Vaginal hemorrhage with undetermined etiology

Ages: 35 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2014-09-09 (Actual); Primary Completion 2022-10-11 (Actual); Study Completion 2022-10-11 (Actual)

PRIMARY OUTCOMES:
Postoperative digestive function | 24 months
  Composite variable: patient considering that digestive function is normal AND the Knowles-Eccersley-Scott-Symptom Questionnaire (KESS score) <7 AND the Gastrointestinal Quality of Life Index (GIQLI) score >100.

SECONDARY OUTCOMES:
Unfavorable digestive functional outcome | 24 months
  Presence of severe constipation (<1 stool/5D), increased frequency of daily bowel movements (>=3 stools/D), anal incontinence, postoperative dysuria

OTHER OUTCOMES:
Assessment of digestive function | 24 months
  The Knowles-Eccersley-Scott-Symptom Questionnaire (KESS score), the Gastrointestinal Quality of Life Index (GIQLI), Wexner score of anal continence, Bristol stools score.

CONTACTS AND LOCATIONS:
Locations (11):
- France (11):
  - CHU d'AMIENS, Amiens
  - Service de Gynécologie, Obstétrique et Médecine de la Reproduction CHU de CLERMONT-FERRAND Hôpital ESTAING 1 place Lucie Aubrac, Clermont-Ferrand
  - CHU de DIJON, Dijon
  - Hôpital du CHESNAY, Le Chesnay
  - Service de Gynécologie-Obstétrique AP-HP Hôpital du KREMLIN BICETRE, Le Kremlin-Bicêtre
  - Clinique Gynécologique CHRU de LILLE, Lille
  - Service de Gynécologie-Obstétrique CHU de NIMES, Nîmes
  - Hôpital de TENON, Paris
  - Chi Poissy-St Germain En Laye Poissy, Poissy
  - Clinique Gynécologique et Obstétricale, Rouen
  - CHU de STRASBOURG STRASBOURG, Strasbourg